CLINICAL TRIAL: NCT03621059
Title: Behavioral Therapy for Children and Adolescents With Tourette Syndrome: A Randomized Controlled Trial in Taiwan
Brief Title: Behavioral Therapy for Children and Adolescents With Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chang, Hsiu-Ju, professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ju07310520
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; behavior therapy; children and adolescents
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: A collection of behavioral skills named as Comprehensive Behavioral Intervention (CBIT) for Tics had been found to be effective (Piacentini et al., 2010).The major components of CBIT includes psychoeducation of tics, habit reversal training (HRT), function-based interventions, and relaxation training (Piacentini et al., 2010).The HRT consists of several therapeutic activities, including awareness training (i.e., observing the premonitory urge or other signs preceding the occurrence of a tic), competing response training (i.e., engaging in a voluntary behavior that is physically incompatible with the tic to manage the premonitory urge), self-monitoring of tics and relaxation training (Himle et al., 2006).
Who Masked: Participant
Masking Description: Eligible children were randomly assigned by sealed envelope to either intervention or control group. Several methods were used to maintain the treatment blindly, including segregation of assessment and treatment staff and instructions to children and parents to avoid discussions of treatment assignment with the independent evaluators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Therapy with TS (Experimental): habit reversal training (HRT)
  Interventions: Behavioral: habit reversal training (HRT)
- observational (No Intervention): observational and usual care Pyridoxine(50mg)

INTERVENTIONS:
Behavioral: habit reversal training (HRT) — The intervention group received 4 sessions during 3months of behavior intervention and then, were reassessed at 3 and 6 months following treatment.
  Pyridoxine(50mg)
  Arms: Behavioral Therapy with TS

SUMMARY:
Tourette Syndrome (TS) is a common neuropsychiatric disorder in childhood and adolescence, and often comorbid with psychiatric comorbidity. Antipsychotic medications are usually the first choices, but may associate with adverse effects. Behavioral intervention for TS has been shown to be an effective treatment for children and adolescents, yet have not been performed and evaluated using control trails in Taiwan.

DETAILED DESCRIPTION:
TS is a common neuropsychiatric disorder in childhood and adolescence, and often comorbid with psychiatric comorbidity. Antipsychotic medications are usually the first choices, but may associate with adverse effects. Behavioral intervention for TS has been shown to be an effective treatment for children and adolescents, yet have not been performed and evaluated using control trails in Taiwan. This study therefore was to evaluate the efficacy of a comprehensive behavioral intervention therapy on improving tics and tic-related impairment for children and adolescents with Tourette syndrome.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Diagnostic Criteria For Tourette Syndrome
* Patients aged from 6-15 years who were diagnosed with TS or CTD,
* Never received any pharmacological treatment
* Ability to understand the study purpose and/or provide consent for participation independently and via a caregiver serving as a proxy

Exclusion Criteria:

* Have been diagnosed with another mental illness,
* Had no physical or medical condition,
* Had been received CBIT or cognitive behavior therapy before.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Eefficacy of a behavioral therapy on improving tics with Tourette syndrome | at 3rd month and 6rd months following treatment.
  Behavioral intervention group led to a significantly greater decrease in total motor score on the Yale Global Tic Severity Scale .The gold-standard measure of tic severity in TS, the YGTSS is a clinician-completed measure consisting of a tic symptom checklist, motor and vocal tic severity ratings, and a global tic impairment rating. To ascertain tic severity ratings, the examiner rates five different dimensions of tic severity each on a 0-5 scale: tic number, frequency, duration, intensity, and complexity. Each of the dimensions is scored separately for motor and vocal tics to produce motor and vocal tic subscale scores (range 0-25). These subscales are then combined to produce a total tic severity score (range 0-50), with higher numbers indicating more severe tics. The YGTSS has demonstrated acceptable internal consistency and acceptable convergent and divergent validity).

CONTACTS AND LOCATIONS:
Overall Officials: hsiu-ju Chang, PHD, Principal Investigator — Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bitsko RH, Holbrook JR, Visser SN, Mink JW, Zinner SH, Ghandour RM, Blumberg SJ. A national profile of Tourette syndrome, 2011-2012. J Dev Behav Pediatr. 2014 Jun;35(5):317-22. doi: 10.1097/DBP.0000000000000065. PMID 24906033
- [Result] Robertson MM, Eapen V, Cavanna AE. The international prevalence, epidemiology, and clinical phenomenology of Tourette syndrome: a cross-cultural perspective. J Psychosom Res. 2009 Dec;67(6):475-83. doi: 10.1016/j.jpsychores.2009.07.010. PMID 19913651
- [Result] Wang HS, Kuo MF. Tourette's syndrome in Taiwan: an epidemiological study of tic disorders in an elementary school at Taipei County. Brain Dev. 2003 Dec;25 Suppl 1:S29-31. doi: 10.1016/s0387-7604(03)90005-2. PMID 14980369
- [Result] Chou IC, Lin HC, Lin CC, Sung FC, Kao CH. Tourette syndrome and risk of depression: a population-based cohort study in Taiwan. J Dev Behav Pediatr. 2013 Apr;34(3):181-5. doi: 10.1097/DBP.0b013e3182829f2b. PMID 23572168
- [Result] King RA, Scahill L. Emotional and behavioral difficulties associated with Tourette syndrome. Adv Neurol. 2001;85:79-88. No abstract available. PMID 11530448
- [Result] Robertson MM, Banerjee S, Eapen V, Fox-Hiley P. Obsessive compulsive behaviour and depressive symptoms in young people with Tourette syndrome. A controlled study. Eur Child Adolesc Psychiatry. 2002 Dec;11(6):261-5. doi: 10.1007/s00787-002-0301-3. PMID 12541004
- [Result] Rizzo R, Gulisano M, Pellico A, Cali PV, Curatolo P. Tourette syndrome and comorbid conditions: a spectrum of different severities and complexities. J Child Neurol. 2014 Oct;29(10):1383-9. doi: 10.1177/0883073814534317. Epub 2014 May 14. PMID 24832397
- [Result] Leckman JF, Zhang H, Vitale A, Lahnin F, Lynch K, Bondi C, Kim YS, Peterson BS. Course of tic severity in Tourette syndrome: the first two decades. Pediatrics. 1998 Jul;102(1 Pt 1):14-9. doi: 10.1542/peds.102.1.14. PMID 9651407
- [Result] Elstner K, Selai CE, Trimble MR, Robertson MM. Quality of Life (QOL) of patients with Gilles de la Tourette's syndrome. Acta Psychiatr Scand. 2001 Jan;103(1):52-9. doi: 10.1034/j.1600-0447.2001.00147.x. PMID 11202129
- [Result] Shprecher D, Kurlan R. The management of tics. Mov Disord. 2009 Jan 15;24(1):15-24. doi: 10.1002/mds.22378. PMID 19170198
- [Result] Muller-Vahl KR, Buddensiek N, Geomelas M, Emrich HM. The influence of different food and drink on tics in Tourette syndrome. Acta Paediatr. 2008 Apr;97(4):442-6. doi: 10.1111/j.1651-2227.2008.00675.x. Epub 2008 Feb 27. PMID 18307557
- [Result] Garcia-Lopez R, Perea-Milla E, Garcia CR, Rivas-Ruiz F, Romero-Gonzalez J, Moreno JL, Faus V, Aguas Gdel C, Diaz JC. New therapeutic approach to Tourette Syndrome in children based on a randomized placebo-controlled double-blind phase IV study of the effectiveness and safety of magnesium and vitamin B6. Trials. 2009 Mar 10;10:16. doi: 10.1186/1745-6215-10-16. PMID 19284553
- [Result] Scahill L, Erenberg G, Berlin CM Jr, Budman C, Coffey BJ, Jankovic J, Kiessling L, King RA, Kurlan R, Lang A, Mink J, Murphy T, Zinner S, Walkup J; Tourette Syndrome Association Medical Advisory Board: Practice Committee. Contemporary assessment and pharmacotherapy of Tourette syndrome. NeuroRx. 2006 Apr;3(2):192-206. doi: 10.1016/j.nurx.2006.01.009. PMID 16554257
- [Result] Roessner V, Plessen KJ, Rothenberger A, Ludolph AG, Rizzo R, Skov L, Strand G, Stern JS, Termine C, Hoekstra PJ; ESSTS Guidelines Group. European clinical guidelines for Tourette syndrome and other tic disorders. Part II: pharmacological treatment. Eur Child Adolesc Psychiatry. 2011 Apr;20(4):173-96. doi: 10.1007/s00787-011-0163-7. PMID 21445724
- [Result] Bruggeman R, van der Linden C, Buitelaar JK, Gericke GS, Hawkridge SM, Temlett JA. Risperidone versus pimozide in Tourette's disorder: a comparative double-blind parallel-group study. J Clin Psychiatry. 2001 Jan;62(1):50-6. doi: 10.4088/jcp.v62n0111. PMID 11235929
- [Result] Sallee FR, Gilbert DL, Vinks AA, Miceli JJ, Robarge L, Wilner K. Pharmacodynamics of ziprasidone in children and adolescents: impact on dopamine transmission. J Am Acad Child Adolesc Psychiatry. 2003 Aug;42(8):902-7. doi: 10.1097/01.CHI.0000046897.27264.46. PMID 12874491
- [Result] Bressan RA, Jones HM, Pilowsky LS. Atypical antipsychotic drugs and tardive dyskinesia: relevance of D2 receptor affinity. J Psychopharmacol. 2004 Mar;18(1):124-7. doi: 10.1177/0269881104040251. PMID 15107196
- [Result] Gaffney GR, Perry PJ, Lund BC, Bever-Stille KA, Arndt S, Kuperman S. Risperidone versus clonidine in the treatment of children and adolescents with Tourette's syndrome. J Am Acad Child Adolesc Psychiatry. 2002 Mar;41(3):330-6. doi: 10.1097/00004583-200203000-00013. PMID 11886028
- [Result] Du YS, Li HF, Vance A, Zhong YQ, Jiao FY, Wang HM, Wang MJ, Su LY, Yu DL, Ma SW, Wu JB. Randomized double-blind multicentre placebo-controlled clinical trial of the clonidine adhesive patch for the treatment of tic disorders. Aust N Z J Psychiatry. 2008 Sep;42(9):807-13. doi: 10.1080/00048670802277222. PMID 18696285
- [Result] Ho CS, Chen HJ, Chiu NC, Shen EY, Lue HC. Short-term sulpiride treatment of children and adolescents with Tourette syndrome or chronic tic disorder. J Formos Med Assoc. 2009 Oct;108(10):788-93. doi: 10.1016/S0929-6646(09)60406-X. PMID 19864199
- [Result] Kim DD, Warburton DER, Wu N, Barr AM, Honer WG, Procyshyn RM. Effects of physical activity on the symptoms of Tourette syndrome: A systematic review. Eur Psychiatry. 2018 Feb;48:13-19. doi: 10.1016/j.eurpsy.2017.11.002. Epub 2018 Jan 10. PMID 29331594
- [Result] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Result] Dutta N, Cavanna AE. The effectiveness of habit reversal therapy in the treatment of Tourette syndrome and other chronic tic disorders: a systematic review. Funct Neurol. 2013 Jan-Mar;28(1):7-12. PMID 23731910
- [Result] Himle MB, Woods DW, Piacentini JC, Walkup JT. Brief review of habit reversal training for Tourette syndrome. J Child Neurol. 2006 Aug;21(8):719-25. doi: 10.1177/08830738060210080101. PMID 16970874
- [Result] Azrin NH, Nunn RG. Habit-reversal: a method of eliminating nervous habits and tics. Behav Res Ther. 1973 Nov;11(4):619-28. doi: 10.1016/0005-7967(73)90119-8. No abstract available. PMID 4777653
- [Result] Woods DW, Miltenberger RG. Habit reversal: a review of applications and variations. J Behav Ther Exp Psychiatry. 1995 Jun;26(2):123-31. doi: 10.1016/0005-7916(95)00009-o. PMID 7593685
- [Result] Watson TS, Sterling HE. Brief functional analysis and treatment of a vocal tic. J Appl Behav Anal. 1998 Fall;31(3):471-4. doi: 10.1901/jaba.1998.31-471. PMID 9757584
- [Result] Blount TH, Lockhart AL, Garcia RV, Raj JJ, Peterson AL. Intensive outpatient comprehensive behavioral intervention for tics: A case series. World J Clin Cases. 2014 Oct 16;2(10):569-77. doi: 10.12998/wjcc.v2.i10.569. PMID 25325069
- [Result] Deckersbach T, Rauch S, Buhlmann U, Wilhelm S. Habit reversal versus supportive psychotherapy in Tourette's disorder: a randomized controlled trial and predictors of treatment response. Behav Res Ther. 2006 Aug;44(8):1079-90. doi: 10.1016/j.brat.2005.08.007. Epub 2005 Nov 2. PMID 16259942
- [Result] Wilhelm S, Peterson AL, Piacentini J, Woods DW, Deckersbach T, Sukhodolsky DG, Chang S, Liu H, Dziura J, Walkup JT, Scahill L. Randomized trial of behavior therapy for adults with Tourette syndrome. Arch Gen Psychiatry. 2012 Aug;69(8):795-803. doi: 10.1001/archgenpsychiatry.2011.1528. PMID 22868933
- [Result] Abramovitch A, Reese H, Woods DW, Peterson A, Deckersbach T, Piacentini J, Scahill L, Wilhelm S. Psychometric Properties of a Self-Report Instrument for the Assessment of Tic Severity in Adults With Tic Disorders. Behav Ther. 2015 Nov;46(6):786-96. doi: 10.1016/j.beth.2015.06.002. Epub 2015 Jun 18. PMID 26520221
- [Result] Storch EA, Murphy TK, Geffken GR, Sajid M, Allen P, Roberti JW, Goodman WK. Reliability and validity of the Yale Global Tic Severity Scale. Psychol Assess. 2005 Dec;17(4):486-91. doi: 10.1037/1040-3590.17.4.486. PMID 16393016
- [Result] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Result] Azrin NH, Peterson AL. Habit reversal for the treatment of Tourette syndrome. Behav Res Ther. 1988;26(4):347-51. doi: 10.1016/0005-7967(88)90089-7. No abstract available. PMID 3214400
- [Result] Yates R, Edwards K, King J, Luzon O, Evangeli M, Stark D, McFarlane F, Heyman I, Ince B, Kodric J, Murphy T. Habit reversal training and educational group treatments for children with tourette syndrome: A preliminary randomised controlled trial. Behav Res Ther. 2016 May;80:43-50. doi: 10.1016/j.brat.2016.03.003. Epub 2016 Mar 23. PMID 27037483
- [Result] Rizzo R, Pellico A, Silvestri PR, Chiarotti F, Cardona F. A Randomized Controlled Trial Comparing Behavioral, Educational, and Pharmacological Treatments in Youths With Chronic Tic Disorder or Tourette Syndrome. Front Psychiatry. 2018 Mar 27;9:100. doi: 10.3389/fpsyt.2018.00100. eCollection 2018. PMID 29636706
- [Result] Woods DW, Twohig MP, Flessner CA, Roloff TJ. Treatment of vocal tics in children with Tourette syndrome: investigating the efficacy of habit reversal. J Appl Behav Anal. 2003 Spring;36(1):109-12. doi: 10.1901/jaba.2003.36-109. PMID 12723873